CLINICAL TRIAL: NCT00537823
Title: Effect of Short-duration Preoperative Neoadjuvant Therapy With FOLFOX Based Therapy on Morbidity After Liver Resection for Colorectal Cancer Metastases
Brief Title: Pre- and Post-operative FOLFOX Based Therapy for Patients With Colorectal Cancer With Liver Involvement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0182
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer; Metastases
Keywords: Colorectal Cancer; Metastasis; Neoadjuvant Therapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Bevacizumab; Leucovorin; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 - Wildtype (Experimental): Neoadjuvant therapy
  Week 1
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV Cetuximab 400 mg/m2 IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2/day over 46 hours
  Weeks 2, 4, 6, 8 *Cetuximab 250 mg/m^2 IV weekly
  Weeks 3, 5, 7
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV Cetuximab 400 mg/m^2 IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2/day over 46 hours
  Wait 3-8 weeks after completion of therapy
  Liver resection
  Wait 4 weeks or until clinical status allows
  Adjuvant Therapy
  Week 1, 3, 5, 7, 9, 11, 13, 15
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV Cetuximab 400 mg/m^2 IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2/day over 46 hours
  Weeks 2, 4, 6, 8, 10, 12, 16
  *Cetuximab 250 mg/m^2 IV weekly
  Interventions: Drug: Cetuximab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Fluorouracil
- Arm 2 K-Ras 12/13 codon mutation (Experimental): Neoadjuvant Therapy
  Weeks 1, 3, 5
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV
  * Bevacizumab 5 mg/kg IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2
  Week 7
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2
  Wait 3-8 weeks after completion of therapy
  Liver resection
  Wait 4 weeks or until clinical status allows
  Adjuvant Therapy
  Weeks 1, 3, 5, 9, 11, 13
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV
  * Bevacizumab 5 mg/kg IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2
  Week 7, 15
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2
  Interventions: Drug: Bevacizumab; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Cetuximab
  Other Names: Erbitux
  Arms: Arm 1 - Wildtype
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Arm 2 K-Ras 12/13 codon mutation
Drug: Leucovorin
Drug: Oxaliplatin
Drug: Fluorouracil

SUMMARY:
The purpose of this study is to determine the effect of short-duration pre-operative FOLFOX based therapy on postoperative problems after liver surgery for patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Although early stage, localized colon and rectal cancers are associated with 5 year survival rates of nearly 90%, only a minority of patients present with localized disease. Unfortunately, at the time of their initial presentation, approximately 35% of patients with colon or rectal cancer have metastatic disease. Nearly two thirds of these patients with stage IV disease have evidence of extrahepatic spread and have a median overall survival rate of 8-10 months in the absence of further treatment. Even with the most intensive chemotherapeutic regimens, the median overall survival for these patients ranges from 12 months to 20 months. However, a small subset of patients with stage IV disease has isolated hepatic metastatic disease and can undergo resection. The patients with completely resected liver metastases enjoy a significantly higher overall five-year survival, which is as high as 58% in carefully selected patients. Ten-year overall survival has been reported in 22% of patients. Despite this improvement, the five-year disease-free survival for these patients is at best 35%, with hepatic recurrences occurring in 46%.

The fact that adjuvant chemotherapy improves the three-year survival rate for stage II disease and five-year survival rates for stage III disease implies that it can treat micrometastatic disease in some fraction of patients. Because micrometastatic disease is likely the cause of the high recurrence rate in patients who undergo liver resection, there is a clear biologic rationale for using postoperative adjuvant chemotherapy after liver resection. Although this strategy is a common practice in many centers, no convincing data that this improves survival have been reported. A large randomized phase III trial (EORTC 40983) examining this question is currently ongoing and effect on survival has not yet been reported. Given that systemic chemotherapy after liver resection remains of unproven benefit at the present time, many have wondered if preoperative treatment might have more promise in improving recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* Synchronous or metachronous colorectal metastases
* Technically resectable liver metastases

  * Four or fewer metastases
  * No tumors in porta hepatis
  * Resection of no more than 70% of liver needed
* Medically suitable candidate for major liver resection
* FDG-PET scan without metastatic disease outside the liver

Exclusion Criteria:

* Near-obstructing or obstructing colon lesions in patients in whom combined resection is planned (as delay for preoperative chemotherapy would be medially impossible)
* Treatment with FOLFOX or cetuximab within 12 months
* Treatment with irinotecan within 12 months
* Abnormal liver function (ALT or AST > 5x ULN, bilirubin > 3x ULN)
* Body mass index >/= 35 kg/m² (as the risk for steatohepatitis is increased)
* Renal insufficiency (Cr > 2.5mg/dL)
* Interstitial lung disease (because cetuximab has been rarely associated with development of interstitial lung disease)
* ECOG performance score >/= 3
* Patients unable to give informed consent
* Pregnant patient (as cetuximab is a Class C drug)
* Peripheral neuropathy >/= grade II (as oxaliplatin causes neuropathy to worsen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Linehan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Adam R, Aloia T, Figueras J, Capussotti L, Poston G, Mentha G, Selzner M, and the LiverMetSurvey Scientific Committee. LiverMetSurvey: Analysis of clinicopathologic factors associated with the efficacy of preoperative chemotherapy in 2,122 patients with colorectal liver metastases. Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings Part I. Vol 24, No. 18S (June 20 Supplement), 2006: 3521.
- [Background] Adam R, Avisar E, Ariche A, Giachetti S, Azoulay D, Castaing D, Kunstlinger F, Levi F, Bismuth F. Five-year survival following hepatic resection after neoadjuvant therapy for nonresectable colorectal. Ann Surg Oncol. 2001 May;8(4):347-53. doi: 10.1007/s10434-001-0347-3. PMID 11352309
- [Background] Alberts SR, Horvath WL, Sternfeld WC, Goldberg RM, Mahoney MR, Dakhil SR, Levitt R, Rowland K, Nair S, Sargent DJ, Donohue JH. Oxaliplatin, fluorouracil, and leucovorin for patients with unresectable liver-only metastases from colorectal cancer: a North Central Cancer Treatment Group phase II study. J Clin Oncol. 2005 Dec 20;23(36):9243-9. doi: 10.1200/JCO.2005.07.740. Epub 2005 Oct 17. PMID 16230673
- [Background] Andre T, Boni C, Mounedji-Boudiaf L, Navarro M, Tabernero J, Hickish T, Topham C, Zaninelli M, Clingan P, Bridgewater J, Tabah-Fisch I, de Gramont A; Multicenter International Study of Oxaliplatin/5-Fluorouracil/Leucovorin in the Adjuvant Treatment of Colon Cancer (MOSAIC) Investigators. Oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment for colon cancer. N Engl J Med. 2004 Jun 3;350(23):2343-51. doi: 10.1056/NEJMoa032709. PMID 15175436
- [Background] Badarinath S, Mitchell EP, Jennis A, Graham CD, Hansen VL, Henderson CA, Chen TT, Langer C. Cetuximab plus FOLFOX for colorectal cancer (EXPLORE): Preliminary safety analysis of a randomized phase III trial. Journal of Clinical Oncology, 2004 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 22, No 14S (July 15 Supplement), 2004: 3531.
- [Background] Bilchik AJ, Poston G, Curley SA, Strasberg S, Saltz L, Adam R, Nordlinger B, Rougier P, Rosen LS. Neoadjuvant chemotherapy for metastatic colon cancer: a cautionary note. J Clin Oncol. 2005 Dec 20;23(36):9073-8. doi: 10.1200/JCO.2005.03.2334. No abstract available. PMID 16361615
- [Background] Capussotti L, Muratore A, Ferrero A, Massucco P, Ribero D, Polastri R. Randomized clinical trial of liver resection with and without hepatic pedicle clamping. Br J Surg. 2006 Jun;93(6):685-9. doi: 10.1002/bjs.5301. PMID 16703653
- [Background] Clavien PA, Sanabria JR, Strasberg SM. Proposed classification of complications of surgery with examples of utility in cholecystectomy. Surgery. 1992 May;111(5):518-26. PMID 1598671
- [Background] Colucci G, Giuliani F, Mattioli R, Garufi C, Mallamaci R, Pezzella G, Lopez M, Maiello E. FOLFOX-4 + cetuximab in untreated patients with advanced colorectal cancer. A phase II study of the Gruppo Oncologico dell'Italia Meridionale . Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings Part I. Vol 24, No. 18S (June 20 Supplement), 2006: 3559.
- [Background] Cunningham D, Humblet Y, Siena S, Khayat D, Bleiberg H, Santoro A, Bets D, Mueser M, Harstrick A, Verslype C, Chau I, Van Cutsem E. Cetuximab monotherapy and cetuximab plus irinotecan in irinotecan-refractory metastatic colorectal cancer. N Engl J Med. 2004 Jul 22;351(4):337-45. doi: 10.1056/NEJMoa033025. PMID 15269313
- [Background] Dakhil S, Cosgriff T, Headley D, Badarinath S, International Oncology Network, R. V. Boccia. Cetuximab + FOLFOX6 as first line therapy for metastatic colorectal cancer. Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings Part I. Vol 24, No. 18S, 2006: 3557
- [Background] D'Angelica M, Maddineni S, Fong Y, Martin RC, Cohen MS, Ben-Porat L, Gonen M, DeMatteo RP, Blumgart LH, Jarnagin WR. Optimal abdominal incision for partial hepatectomy: increased late complications with Mercedes-type incisions compared to extended right subcostal incisions. World J Surg. 2006 Mar;30(3):410-8. doi: 10.1007/s00268-005-0183-x. PMID 16467983
- [Background] Delaunoit T, Alberts SR, Sargent DJ, Green E, Goldberg RM, Krook J, Fuchs C, Ramanathan RK, Williamson SK, Morton RF, Findlay BP. Chemotherapy permits resection of metastatic colorectal cancer: experience from Intergroup N9741. Ann Oncol. 2005 Mar;16(3):425-9. doi: 10.1093/annonc/mdi092. Epub 2005 Jan 27. PMID 15677624
- [Background] Díaz Rubio E, JTabernero J, van Cutsem E, Cervantes A, André T, Humblet Y, Soulié P, Corretgé S, Kisker O,de Gramont A. Cetuximab in combination with oxaliplatin/5-fluorouracil (5-FU)/folinic acid (FA) (FOLFOX-4) in the first-line treatment of patients with epidermal growth factor receptor (EGFR)-expressing metastatic colorectal cancer: An international phase II study. Journal of Clinical Oncology, 2005 ASCO Annual Meeting Proceedings. Vol 23, No. 16S, Part I of II (June 1 Supplement), 2005: 3535.
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Ellis LM, Curley SA, Grothey A. Surgical resection after downsizing of colorectal liver metastasis in the era of bevacizumab. J Clin Oncol. 2005 Aug 1;23(22):4853-5. doi: 10.1200/JCO.2005.23.754. No abstract available. PMID 16051943
- [Background] Fausto N, Campbell JS, Riehle KJ. Liver regeneration. Hepatology. 2006 Feb;43(2 Suppl 1):S45-53. doi: 10.1002/hep.20969. PMID 16447274
- [Background] Fernandez FG, Drebin JA, Linehan DC, Dehdashti F, Siegel BA, Strasberg SM. Five-year survival after resection of hepatic metastases from colorectal cancer in patients screened by positron emission tomography with F-18 fluorodeoxyglucose (FDG-PET). Ann Surg. 2004 Sep;240(3):438-47; discussion 447-50. doi: 10.1097/01.sla.0000138076.72547.b1. PMID 15319715
- [Background] Fernandez FG, Ritter J, Goodwin JW, Linehan DC, Hawkins WG, Strasberg SM. Effect of steatohepatitis associated with irinotecan or oxaliplatin pretreatment on resectability of hepatic colorectal metastases. J Am Coll Surg. 2005 Jun;200(6):845-53. doi: 10.1016/j.jamcollsurg.2005.01.024. PMID 15922194
- [Background] Finkelstein SE, Fernandez FG, Dehdashti F, Siegel BA, Hawkins WG, Linehan DC, Strasberg SM. Unique site- and time-specific patterns of recurrence following resection of colorectal carcinoma hepatic metastases in patients staged by FDG-PET. J Hepatobiliary Pancreat Surg. 2008;15(5):483-7. doi: 10.1007/s00534-007-1237-2. Epub 2008 Oct 4. PMID 18836801
- [Background] Gruenberger T, Sorbye H, Debois M, Bethe U, Primrose J, Rougier P, Jaeck D, Finch-Jones M, Van Cutsem E, Nordlinger B. Tumor response to pre-operative chemotherapy (CT) with FOLFOX-4 for resectable colorectal cancer liver metastases (LM). Interim results of EORTC Intergroup randomized phase III study 40983. Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings Part I. Vol 24, No. 18S (June 20 Supplement), 2006: 3500.
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Ibrahim S, Chen CL, Wang CC, Wang SH, Lin CC, Liu YW, Yang CH, Yong CC, Concejero A, Cheng YF. Liver regeneration and splenic enlargement in donors after living-donor liver transplantation. World J Surg. 2005 Dec;29(12):1658-66. doi: 10.1007/s00268-005-0101-2. PMID 16311869
- [Background] Jennis A , J. Polikoff, E. Mitchell, S. Badarinath, C. Graham, T. Chen, T. Gustafson, C. Langer Erbitux (Cetuximab) Plus FOLFOX for Colorectal Cancer (EXPLORE): Preliminary efficacy analysis of a randomized phase III trial. Journal of Clinical Oncology, 2005 ASCO Annual Meeting Proceedings. Vol 23, No. 16S, Part I of II (June 1 Supplement), 2005: 3574
- [Background] Karoui M, Penna C, Amin-Hashem M, Mitry E, Benoist S, Franc B, Rougier P, Nordlinger B. Influence of preoperative chemotherapy on the risk of major hepatectomy for colorectal liver metastases. Ann Surg. 2006 Jan;243(1):1-7. doi: 10.1097/01.sla.0000193603.26265.c3. PMID 16371728
- [Background] Koniaris LG, McKillop IH, Schwartz SI, Zimmers TA. Liver regeneration. J Am Coll Surg. 2003 Oct;197(4):634-59. doi: 10.1016/S1072-7515(03)00374-0. No abstract available. PMID 14522336
- [Background] Lorenz M, Staib-Sebler E, Gog C, Proschek D, Jauch KW, Ridwelski K, Hohenberger W, Gassel HJ, Lehmann U, Vestweber KH, Padberg W, Zamzow K, Muller HH. Prospective pilot study of neoadjuvant chemotherapy with 5-fluorouracil, folinic acid and oxaliplatin in resectable liver metastases of colorectal cancer. Analysis of 42 neoadjuvant chemotherapies. Zentralbl Chir. 2003 Feb;128(2):87-94. doi: 10.1055/s-2003-37760. PMID 12632273
- [Background] Moertel CG, Fleming TR, Macdonald JS, Haller DG, Laurie JA, Goodman PJ, Ungerleider JS, Emerson WA, Tormey DC, Glick JH, et al. Levamisole and fluorouracil for adjuvant therapy of resected colon carcinoma. N Engl J Med. 1990 Feb 8;322(6):352-8. doi: 10.1056/NEJM199002083220602. PMID 2300087
- [Background] Nordlinger B, Sorbye H, Debois M, Praet M, Glimelius B, Poston GJ, P. Schlag M, Walpole ET, Bechstein W, Gruenberger T. Feasibility and risks of pre-operati ve chemotherapy (CT) with Folfox 4 and surgery for resectable colorectal cancer liver metastases (LM). Interim results of the EORTC Intergroup randomized phase III study 40983. Journal of Clinical Oncology, 2005 ASCO Annual Meeting Proceedings. Vol 23, No. 16S, Part I of II (June 1 Supplement), 2005: 3528.
- [Background] Portier G, Rougier P, Milan C et al. Adjuvant systemic chemotherapy using 5-fluorouracil and folinic acid after resection of liver metastases from colorectal origin. Results of an intergroup phase III study (trial FFCD-ACHBTH-AURC 9002). Proc Am Soc Clin Oncol (2002); 20:528 (abstr).
- [Background] Reddy GK. The addition of bevacizumab to FOLFOX4 prolongs survival in relapsed colorectal cancer: interim data from the ECOG 3200 trial. Clin Colorectal Cancer. 2005 Jan;4(5):300-1. doi: 10.1016/s1533-0028(11)70131-1. No abstract available. PMID 15663832
- [Background] Scappaticci FA, Fehrenbacher L, Cartwright T, Hainsworth JD, Heim W, Berlin J, Kabbinavar F, Novotny W, Sarkar S, Hurwitz H. Surgical wound healing complications in metastatic colorectal cancer patients treated with bevacizumab. J Surg Oncol. 2005 Sep 1;91(3):173-80. doi: 10.1002/jso.20301. PMID 16118771
- [Background] Schemmer P, Friess H, Hinz U, Mehrabi A, Kraus TW, Z'graggen K, Schmidt J, Uhl W, Buchler MW. Stapler hepatectomy is a safe dissection technique: analysis of 300 patients. World J Surg. 2006 Mar;30(3):419-30. doi: 10.1007/s00268-005-0192-9. PMID 16467982
- [Background] Shah SA, Haddad R, Al-Sukhni W, Kim RD, Greig PD, Grant DR, Taylor BR, Langer B, Gallinger S, Wei AC. Surgical resection of hepatic and pulmonary metastases from colorectal carcinoma. J Am Coll Surg. 2006 Mar;202(3):468-75. doi: 10.1016/j.jamcollsurg.2005.11.008. Epub 2006 Jan 18. PMID 16500252
- [Background] Tabernero JM, Van Cutsem E, Sastre J, Cervantes A, Van Laethem JL, Humblet Y, Soulié P, Corretgé S, Mueser M, De Gramont A; Vall d'Hebron. An international phase II study of cetuximab in combination with oxaliplatin/5-fluorouracil (5-FU)/folinic acid (FA) (FOLFOX-4) in the first-line treatment of patients with metastatic colorectal cancer (CRC) expressing Epidermal Growth Factor Receptor (EGFR). Preliminary results. Journal of Clinical Oncology, 2004 ASCO Annual Meeting Proceedings (Post-Meeting Edition). Vol 22, No 14S (July 15 Supplement), 2004: 3512.
- [Background] Taieb J, Artru P, Paye F, Louvet C, Perez N, Andre T, Gayet B, Hebbar M, Goebel FM, Tournigand C, Parc R, de Gramont A. Intensive systemic chemotherapy combined with surgery for metastatic colorectal cancer: results of a phase II study. J Clin Oncol. 2005 Jan 20;23(3):502-9. doi: 10.1200/JCO.2005.05.082. PMID 15659495
- [Background] Tanaka K, Adam R, Shimada H, Azoulay D, Levi F, Bismuth H. Role of neoadjuvant chemotherapy in the treatment of multiple colorectal metastases to the liver. Br J Surg. 2003 Aug;90(8):963-9. doi: 10.1002/bjs.4160. PMID 12905549
- [Background] Vauthey JN, Pawlik TM, Ribero D, Wu TT, Zorzi D, Hoff PM, Xiong HQ, Eng C, Lauwers GY, Mino-Kenudson M, Risio M, Muratore A, Capussotti L, Curley SA, Abdalla EK. Chemotherapy regimen predicts steatohepatitis and an increase in 90-day mortality after surgery for hepatic colorectal metastases. J Clin Oncol. 2006 May 1;24(13):2065-72. doi: 10.1200/JCO.2005.05.3074. PMID 16648507
- [Background] Venook A, Niedzwiecki D, Hollis D, Sutherland S, Goldberg R, Alberts S, Benson A, Wade J, Schilsky R, Mayer R. Phase III study of irinotecan/5FU/LV (FOLFIRI) or oxaliplatin/5FU/LV (FOLFOX) ± cetuximab for patients with untreated metastatic adenocarcinoma of the colon or rectum (MCRC): CALGB 80203 preliminary results. Journal of Clinical Oncology, 2006 ASCO Annual Meeting Proceedings Part I. Vol 24, No. 18S (June 20 Supplement), 2006: 3509.
- [Background] Wei AC, Greig PD, Grant D, Taylor B, Langer B, Gallinger S. Survival after hepatic resection for colorectal metastases: a 10-year experience. Ann Surg Oncol. 2006 May;13(5):668-76. doi: 10.1245/ASO.2006.05.039. Epub 2006 Mar 10. PMID 16523369
- [Background] Wolmark N, Wieand S, Kuebler JP, Colangelo L, and Smith RE. A phase III trial comparing FULV to FULV + oxaliplatin in stage II or III carcinoma of the colon: Results of NSABP Protocol C-07. ASCO Meeting Abstracts 2005 23.
- [Background] Yedibela S, Elad L, Wein A, Dimmler A, Merkel S, Hohenberger W, Meyer T. Neoadjuvant chemotherapy does not increase postoperative complication rate after resection of colorectal liver metastases. Eur J Surg Oncol. 2005 Mar;31(2):141-6. doi: 10.1016/j.ejso.2004.07.030. PMID 15698729
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 06/06/2007 and closed to participants enrollment on 11/03/2009.
Groups:
- Arm 1 - Wildtype: Neoadjuvant therapy
  Week 1
  * Leucovorin 400 mg/m2 IV
  * Oxaliplatin 85 mg/m2 IV Cetuximab 400 mg/m2 IV
  * 5FU bolus 400 mg/m2
  * 5FU CIVI 1200 mg/m2/day over 46 hours
  Weeks 2, 4, 6, 8 *Cetuximab 250 mg/m2 IV weekly
  Weeks 3, 5, 7
  * Leucovorin 400 mg/m2 IV
  * Oxaliplatin 85 mg/m2 IV Cetuximab 400 mg/m2 IV
  * 5FU bolus 400 mg/m2
  * 5FU CIVI 1200 mg/m2/day over 46 hours
  Wait 3-8 weeks after completion of therapy
  Liver resection
  Wait 4 weeks or until clinical status allows
  Adjuvant Therapy
  Week 1, 3, 5, 7, 9, 11, 13, 15
  * Leucovorin 400 mg/m2 IV
  * Oxaliplatin 85 mg/m2 IV Cetuximab 400 mg/m2 IV
  * 5FU bolus 400 mg/m2
  * 5FU CIVI 1200 mg/m2/day over 46 hours
  Weeks 2, 4, 6, 8, 10, 12, 16
  *Cetuximab 250 mg/m2 IV weekly
- Arm 2 K-Ras 12/13 Codon Mutation: Neoadjuvant Therapy
  Weeks 1, 3, 5
  * Leucovorin 400 mg/m2 IV
  * Oxaliplatin 85 mg/m2 IV
  * Bevacizumab 5 mg/kg IV
  * 5FU bolus 400 mg/m2
  * 5FU CIVI 1200 mg/m2
  Week 7
  * Leucovorin 400 mg/m2 IV
  * Oxaliplatin 85 mg/m2 IV
  * 5FU bolus 400 mg/m2
  * 5FU CIVI 1200 mg/m2
  Wait 3-8 weeks after completion of therapy
  Liver resection
  Wait 4 weeks or until clinical status allows
  Adjuvant Therapy
  Weeks 1, 3, 5, 9, 11, 13
  * Leucovorin 400 mg/m2 IV
  * Oxaliplatin 85 mg/m2 IV
  * Bevacizumab 5 mg/kg IV
  * 5FU bolus 400 mg/m2
  * 5FU CIVI 1200 mg/m2
  Week 7, 15
  * Leucovorin 400 mg/m2 IV
  * Oxaliplatin 85 mg/m2 IV
  * 5FU bolus 400 mg/m2
  * 5FU CIVI 1200 mg/m2
Period: Overall Study
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Started | 7 | 2
Completed | 5 | 2
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 70] | 62 [47 to 77] | 62 [44 to 77]
Gender [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Complication Rate
Description: Fraction of patients with any grade of complication I-V
Time Frame: 30 days following surgery
Population: 4 participants did not have surgery.
Measure: Number; unit: percentage of participants
Groups:
- Arm 1 - Wildtype: Neoadjuvant therapy
  Week 1
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV Cetuximab 400 mg/m^2 IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2/day over 46 hours
  Weeks 2, 4, 6, 8 *Cetuximab 250 mg/m^2 IV weekly
  Weeks 3, 5, 7
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV Cetuximab 400 mg/m^2 IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2/day over 46 hours
  Wait 3-8 weeks after completion of therapy
  Liver resection
  Wait 4 weeks or until clinical status allows
  Adjuvant Therapy
  Week 1, 3, 5, 7, 9, 11, 13, 15
  * Leucovorin 400 mg/m^2 IV
  * Oxaliplatin 85 mg/m^2 IV Cetuximab 400 mg/m^2 IV
  * 5FU bolus 400 mg/m^2
  * 5FU CIVI 1200 mg/m^2/day over 46 hours
  Weeks 2, 4, 6, 8, 10, 12, 16
  *Cetuximab 250 mg/m^2 IV weekly
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 4 | 1
percentage of participants | 25 | 0

2. Primary Outcome: Major Postoperative Complication Rate
Description: Fraction of patients with any complication grades IV and V
Time Frame: 30 days following surgery
Population: 4 participants did not have surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 4 | 1
percentage of participants | 25 | 0

3. Primary Outcome: All-cause Mortality
Time Frame: 30 days following surgery
Population: 4 participants did not have surgery.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 4 | 1
participants | 0 | 0

4. Secondary Outcome: Postoperative Recurrence Patterns
Description: Liver only vs distant disease
Time Frame: Up to 5 years
Population: 7 participants were not evaluable. 4 participants did not have surgery (3 in Arm 1, 1 in Arm 2). 1 participant had surgery but was not resectable (Arm 1) . 1 participant developed another primary cancer (Arm 1). 1 participant died before recurrence from hepatic failure (Arm 1).
Measure: Number; unit: participants
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 1 | 1
participants
  Liver only | 0 | 0
  Distant disease | 1 | 0

5. Secondary Outcome: Histologic Hepatic Toxicity at Surgery
Time Frame: Time of surgery (approximately 11-16 weeks)
Population: 4 participants did not have surgery.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 4 | 1
participants
  Not reported on pathology report | 1 | 0
  Mild | 1 | 0
  Aborted surgery | 1 | 0
  None | 1 | 1

6. Secondary Outcome: Nonalcoholic Steatohepatitis Score (0-3)
Description: * NASH Scoring
    * Steatosis **<5% = 0
      **5-33%=1
      **>33-66%=2
      **>66%=3
    * Lobular inflammation
      **No foci=0
      **<2 foci per x 200 field=1
      **2-4 foci per x 200 field=2
      **>4 foci per x 200 field=3
    * Hepatocellular ballooning **None=0 **Few balloon cells = 1 **Many cells/prominent ballooning=2
Time Frame: Time of surgery (approximately 11-16 weeks)
Population: 4 participants did not have surgery and are not included in this outcome measure.
  The study pathologist left the university early prior to completion of study pathology for this study.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 4 | 1
participants
  Not reported on pathology report | 3 | 0
  Aborted surgery | 1 | 0
  Score 0 | 0 | 1

7. Secondary Outcome: Liver Injury Scale Score (0-27)
Time Frame: Time of surgery (approximately 11-16 weeks)
Population: Data was not collected for this outcome measure as the study pathologist left the institution early prior to study closure.
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Effect of Preoperative Chemotherapy on Tumor Size
Description: Number of participants whose tumor size decreased from baseline to completion of preoperative chemotherapy.
Time Frame: Upon completion of neoadjuvant chemotherapy (approximately 2 months)
Population: 2 participants did not have the CT scan prior to surgery as both did not complete preoperative chemotherapy due to adverse skin reactions to cetuximab.
Measure: Number; unit: participants
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 5 | 2
participants | 4 | 2

9. Secondary Outcome: Change in Tumor Size From Pretreatment to Preoperative CT Scan
Description: -Compare total longest diameter from baseline to preoperative CT scan.
Time Frame: Completion of neoadjuvant therapy (approximately 8 weeks)
Population: as for outcome 8
Measure: Median (Full Range); unit: percentage of change of longest diameter
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Number analyzed (Participants) | 5 | 2
percentage of change of longest diameter | -23.8 [-71.7 to -0.7] | -14.3 [-28.0 to 2.1]

ADVERSE EVENTS:
Arm/Group | Arm 1 - Wildtype | Arm 2 K-Ras 12/13 Codon Mutation
Serious Adverse Events (participants affected / at risk) | 4/7 | 0/2
Other Adverse Events (participants affected / at risk) | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Wildtype (N=7) | Arm 2 K-Ras 12/13 Codon Mutation (N=2)
Hyperbilirubinemia (Investigations) | 2 | 0
Febrile neutropenia (Infections and infestations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0
Death NOS (Hepatobiliary disorders) | 1 | 0 — Liver dysfunction failure (cholestatic jaundice)
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Wildtype (N=7) | Arm 2 K-Ras 12/13 Codon Mutation (N=2)
Seasonal allergies (Immune system disorders) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 6 | 2
Leukocytes (Investigations) | 7 | 2
Lymphopenia (Investigations) | 6 | 2
Neutrophils (Investigations) | 6 | 2
Platelets (Investigations) | 6 | 2
INR (Investigations) | 3 | 2
PTT (Investigations) | 2 | 2
Fatigue (Investigations) | 6 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 2
Diarrhea (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 4 | 2
Resp-bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection grade 1/2 normal ANC - general (wound) (Infections and infestations) | 0 | 1
Infection grade 1/2 normal ANC - pulmonary (sinus) (Infections and infestations) | 0 | 1
Infection grade 1/2 normal ANC - pulmonary (up airway) (Infections and infestations) | 0 | 1
Albumin, serum-low (Metabolism and nutrition disorders) | 4 | 2
Alkaline phosphatase (Investigations) | 4 | 2
ALT (Investigations) | 5 | 2
AST (Investigations) | 5 | 2
Creatinine (Investigations) | 0 | 1
GGT (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Neuropathy - sensory (Nervous system disorders) | 4 | 2
Pain - GI (Abdomen NOS) (Gastrointestinal disorders) | 0 | 1
Pain - Pulmonary (Throat) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Decreased urination (Renal and urinary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0
Pain - Musculoskeletal (Back) (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain - Musculoskeletal (Limb) (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain - Neurology (Headache) (Nervous system disorders) | 0 | 1
Pain - Other (Liver pain) (Hepatobiliary disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Elevated PT (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Rigors/chills (Investigations) | 2 | 0
Sweating (Investigations) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 0
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 | 0
Rash: hand-foot reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Digestive problems (Gastrointestinal disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0
Mucositis (oral cavity) (Gastrointestinal disorders) | 2 | 0
Mucositis (stomach) (Gastrointestinal disorders) | 1 | 0
Hemorrhage (resp-nose) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Liver dysfunction/failure (Hepatobiliary disorders) | 2 | 0
Febrile neutropenia (Infections and infestations) | 1 | 0
Slight puffiness in right upper lip (Investigations) | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Edema: limb (Investigations) | 1 | 0
Bilirubin (Investigations) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0
Muscle weakness - whole body (Musculoskeletal and connective tissue disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Neuropathy (motor) (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes